CLINICAL TRIAL: NCT04239339
Title: Serotonergic Modulation of Cognition, Emotion and Brain Activation in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Cambridge (Other); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Professor Barbara Jacquelyn Sahakian, Professor, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-18038352
Record Dates: First submitted 2020-01-13; First posted 2020-01-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Serotonin; Cognition; Emotion; Neural Activation
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): The placebo control group will be administered the exact same procedure as the intervention group, the only difference being that this group will be administered a placebo pill.
  Interventions: Drug: Placebo
- Intervention Group (Experimental): The intervention group will be administered 20mg of Escitalopram daily for approximately 3 weeks.
  Interventions: Drug: Escitalopram 20 mg

INTERVENTIONS:
Drug: Escitalopram 20 mg — 20mg daily for approximately 3 weeks.
  Arms: Intervention Group
Drug: Placebo — Placebo daily for approximately 3 weeks.
  Arms: Control Group

SUMMARY:
The aim of this project is:

* To apply a pharmacological tool of selective serotonin (5-hydroxytryptamine, 5-HT system) reuptake inhibition in healthy humans. Specifically:
* To investigate how sub-chronic administration of 20 mg of escitalopram affects cognitive performance ('cold' cognition) and social-emotional functioning ('hot' cognition) compared with placebo; and
* To investigate how sub-chronic administration of 20 mg of escitalopram affects functional brain activation during a paradigm of reinforcement learning following drug administration compared with placebo, and how activation relates to cognitive performance and social-emotional functioning.

DETAILED DESCRIPTION:
The aim of this project is:

* To apply a pharmacological tool of selective serotonin (5-hydroxytryptamine, 5-HT system) reuptake inhibition in healthy humans. Specifically:
* To investigate how sub-chronic administration of 20 mg of escitalopram affects cognitive performance ('cold' cognition) and social-emotional functioning ('hot' cognition) compared with placebo; and
* To investigate how sub-chronic administration of 20 mg of escitalopram affects functional brain activation during a paradigm of reinforcement learning following drug administration compared with placebo, and how activation relates to cognitive performance and social-emotional functioning.

Serotonin is a monoamine neurotransmitter implicated in diverse cognitive and affective brain functions. Serotonin has a significant role in the regulation of cognition and mood, including emotional appraisal, perception and flexible behaviour, with 5-HT receptors found in the cortex, amygdala and hippocampus. The investigators have previously shown that in healthy human experimental studies, acute dietary tryptophan depletion induces 'waiting' impulsivity and impulsive behaviours, impairs goal-directed behaviour and shifts behavioural control toward habitual responding when appetitive, but goal-directed when aversive. Reduced availability of forebrain serotonin has also shown to impair a range of cognitive processes, such as psychomotor processing, episodic memory, attention and executive function. Recently, the research team have shown that using an acute and clinically relevant dose (20 mg) of escitalopram impaired learning and cognitive flexibility, but improved response inhibition in healthy humans, suggesting a dissociation of effects possibly mediated by differential modulation of brain serotonin levels in distinct functional neural circuits.

The investigators now aim to investigate the effects of sub-chronic administration of 20 mg of escitalopram (i.e. three weeks) in healthy volunteers using sophisticated neuropsychological testing (Cambridge Neuropsychological Test Automated Battery and EMOTICOM) and functional magnetic resonance imaging (fMRI). Whereas 'cold' cognition refers to the use of non-emotional processing (e.g. episodic memory; spatial working memory), 'hot' cognition is emotion-laden and used in response to stimuli with affective salience (e.g. decision-making under high levels of risk of uncertainty). It has been suggested that cognitive-emotional effects, such as the re-appraisal and re-evaluation of emotions underlying learning mechanisms, may mediate improvements in mood associated with SSRI treatment. This project will help further the understanding of the role of serotonin in the regulation of cognitive and emotional processes, as well the neural correlates underlying reinforcement learning, in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer (male or female) between 18 and 45 years.

Exclusion Criteria:

* Current or former primary psychiatric disorder (DSM IV Axis I or WHO ICD-10 diagnostic classification).
* Current or previous neurological disease, severe somatic disease, or the consumption of drugs likely to influence the test results.
* Non- fluent in Danish or pronounced visual or auditory impairments.
* Current or past learning disability.
* Pregnancy (females).
* Lactation (females).
* Contraindications for MRI (pacemaker, metal implants, etc.).
* Allergy to the ingredients in the administered drug.
* Abnormal ECG (e.g. prolonged QT syndrome).
* Dizzy when changing from supine to upright position (e.g. postural orthostatic tachycardia syndrome).
* Mild hypotension (blood pressure below 100/70 mmHg) or hypertension (blood pressure above 140/90 mmHg).
* Head injury or concussion resulting in loss of consciousness for more than 2 min.
* Alcohol or drug abuse.
* Drug use other than tobacco and alcohol within the last 30 days.
* Hash > 50 x lifetime.
* Drugs > 10 x lifetime (for each substance).
* Nicotine addiction.
* Current psychoactive medication.
* Severe physical impairments affecting eyesight or motor performance.
* Hamilton-6 depression scale score > 5.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Learning Primary Outcome 1: Mean errors Stage 1 (Learning) - Probability Reversal Learning. | 3 years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Primary Outcome 2: Mean errors Stage 2 (Reversal) - Probability Reversal Learning. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Primary Outcome 3: Learning Rate in Reward Trial - Reinforcement Learning. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Primary Outcome 4: Learning Rate in Punishment Trials - Reinforcement Learning. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Primary Outcome 1: Stop Signal Reaction Time - Interleaved Stop Signal Task/Go-NoGo. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Executive Function Primary Outcome 1: Extra Dimensional Set Errors -3Dimensional Intra/Extra Dimensional Shift. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Reinforcement Behaviour Model | 3 Years
  A model comparison will be conducted to determine the winning model of reinforcement behaviour using one, a combination of, or all these parameters. The winning model will be a single outcome model.
  1. Reward Learning Rate
  2. Punishment Learning Rate
  3. Reinforcement Sensitivity
  4. Stimulus Stickiness
Social Cognition Primary Outcome 1: Proportion of offers accepted - Ultimatum Game | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Social Cognition Primary Outcome 2: Agent Guilt Score - Moral Emotions Task. | 3 Years
  3. Agent Shame Score ---------- Moral Emotions Task Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Social Cognition Primary Outcome 3: Agent Shame Score - Moral Emotions Task. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 1: Affective bias in decreasing condition - EMOTICOM Intensity Morphing. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 2: Affective bias for D' - EMOTICOM Emotion Recognition Task. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 3: Detection threshold decreasing - EMOTICOM Intensity Morphing. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 4: D'Prime for Emotion Recognition - EMOTICOM Emotion Recognition Task. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Biofluids: Serum Escitalopram levels | 3 Years
PET Imaging: Cerebral (particularly hippocampal) presynaptic density, as measured with 11 C-UCB-J-PET. | 3 Years
  Collected in a sub-sample of participants.

SECONDARY OUTCOMES:
Learning Secondary Outcome 1: Stage 1 Reward-Stay/Lose-Shift behaviour - Probability Reversal Learning. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 2: Stage 2 Reward-Stay/ Lose-Shift behaviour - Probability Reversal Learning. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 3: Pre Extra Dimension Set Errors - 3Dimensional Intra/Extra Dimensional Shift. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 4: Proportion of Stays - Sequential Model-Based/Model-Free. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 1: Go reaction time - Interleaved Stop Signal Task/Go-NoGo. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 2: Go omission error rate - Interleaved Stop Signal Task/Go-NoGo. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 3: Go commission error rate - Interleaved Stop Signal Task/Go-NoGo. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 4: No-Go error rate - Interleaved Stop Signal Task/Go-NoGo. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Executive Function Secondary Outcome 1: Total Errors Adjusted - 3Dimensional Intra/Extra Dimensional Shift. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Executive Function Secondary Outcome 2: Strategy Score - CANTAB Spatial Working Memory. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Social Cognition Secondary Outcome 1: Fairness Sensitivity---------- Ultimatum Game | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Secondary Outcome 1: Detection threshold increasing - EMOTICOM Intensity Morphing. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Secondary Outcome 2: Affective bias in increasing condition - EMOTICOM Intensity Morphing. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Secondary Outcome 3: Affective bias for Hit Rate - EMOTICOM Emotion Recognition Task. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Secondary Outcome 4: Hit Rate for Emotion Recognition - EMOTICOM Emotion Recognition Task. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Faces and geometric figure discrimination Outcome 1: Accuracy - Faces fMRI paradigm | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Faces and geometric figure discrimination Outcome 2: Response Speed - Faces fMRI paradigm. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Memory Outcome 1: Total Errors Adj - CANTAB Paired Associates Learning | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Memory Outcome 2: First Trial Memory Score - CANTAB Paired Associates Learning. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Memory Outcome 3: Between Search Errors - CANTAB Spatial Working Memory. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Attention Outcome 1: Target Sensitivity (A') - CANTAB Rapid Visual Processing. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Attention Outcome 2: Latency - CANTAB Rapid Visual Processing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Attention Outcome 3: Probability of False Alarms - CANTAB Rapid Visual Processing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome Outcome 1. Quality of Decision Making - EMOTICOM Cambridge Gamble Task. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome 2: Risk Adjustment - EMOTICOM Cambridge Gamble Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome 3: Overall Proportion Bet - EMOTICOM Cambridge Gamble Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome 4: Deliberation Time - EMOTICOM Cambridge Gamble Task. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Psychomotor Speed Outcome 1: Simple reaction time - CANTAB Reaction Time Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Psychomotor Speed Outcome 2: Five Choice reaction time - CANTAB Reaction Time Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. FDR correction, for multiple comparisons, using the Benjamin Hochberg procedure will be applied to the outcomes within each cognitive domain.
Neural Activations and Correlations - Reinforcement Learning fMRI paradigm | 3 Years
  Imaging outcomes will be FWE corrected using Random Field Theory as implemented in SPM12.
Neural Activations and Correlations - Faces fMRI paradigm | 3 Years
  Imaging outcomes will be FWE corrected using Random Field Theory as implemented in SPM12.
Resting State fMRI | 3 Years
  Imaging outcomes will be FWE corrected using Random Field Theory as implemented in SPM12.
Structural VBM | 3 Years
  Imaging outcomes will be FWE corrected using Random Field Theory as implemented in SPM12.
Diffusion Tensor Imaging | 3 Years
Profile of Mood State Score | 3 Years
Beck Depression Inventory-II Score | 3 Years
State-Trait Anxiety Inventory Scale -State Score | 3 Years
State and Trait Aggression Questionnaire-State Score | 3 Years
Baret Impulsivity Scale-State Score | 3 Years
Visual Analogue Scale Score | 3 Years
Interpersonal Reactivity Index Score | 3 Years
Obsessive- Compulsive Inventory Score | 3 Years
Brief Symptom Checklist Score | 3 Years
Pittsburgh Sleep Quality Index Score | 3 Years

OTHER OUTCOMES:
Emotion Recognition Other Outcome 1: Detection threshold decreasing Happy - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 2: Detection threshold decreasing Sad - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 3: Detection threshold decreasing Anger - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 4: Detection threshold decreasing Fear - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 5: Detection threshold decreasing Disgust - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 6: D' Happy - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 7: D' Sad - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 8: D' Fear - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 9: D' Anger - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Activity Level Score | 3 Years
Behavioural Inhibition/ Behavioural Avoidance Scale Score | 3 Years
The Compulsive Personality Assessment Scale Score | 3 Years
Sexuality Questionnaire Score | 3 Years
Edinburgh Handedness Inventory Score | 3 Years
Revised NEO Personality Questionnaire Score | 3 Years
Family History Assessment Module Score | 3 Years
Positive Life Events Score | 3 Years
Stressful Life Events Score | 3 Years
State and Trait Aggression Questionnaire -Trait Score | 3 Years
Barret Impulsivity Scale-Trait Score | 3 Years
The Penn State Worry Questionnaire- Trait Score | 3 Years
The Penn State Worry Questionnaire- State Score | 3 Years
The Self-Control Scale- Trait Score | 3 Years
The Self-Control Scale- State Score | 3 Years
State- Trait Anxiety Inventory- Trait Score | 3 Years
The Warwick-Edinburgh Mental Well-being Scale -Trait Score | 3 Years
The Warwick-Edinburgh Mental Well-being Scale -State Score | 3 Years
Mindful Attention and Awareness Scale -Trait Score | 3 Years
Mindful Attention and Awareness Scale -State Score | 3 Years
The Intolerance of Uncertainty Scale - Trait Score | 3 Years
The Intolerance of Uncertainty Scale - State Score | 3 Years
Verran Snyder-Halpern (VSH) Sleep Scale Score | 3 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Neurobiology Research Unit, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study all data will be uploaded to the existing CIMBI Database. Researchers may apply for access to the data.
Time Frame: Upon Compeletion of the Study.
Access Criteria: Researchers may apply for access to the data.
URL: https://www.cimbi.dk/

REFERENCES:
- [Background] Homberg JR. Serotonin and decision making processes. Neurosci Biobehav Rev. 2012 Jan;36(1):218-36. doi: 10.1016/j.neubiorev.2011.06.001. Epub 2011 Jun 12. PMID 21693132
- [Background] Meneses A. Are 5-HT(1B/1D) and 5-HT(2A/2B/2C) receptors involved in learning and memory processes? IDrugs. 1999 Aug;2(8):796-801. PMID 16127655
- [Background] Worbe Y, Savulich G, Voon V, Fernandez-Egea E, Robbins TW. Serotonin depletion induces 'waiting impulsivity' on the human four-choice serial reaction time task: cross-species translational significance. Neuropsychopharmacology. 2014 May;39(6):1519-26. doi: 10.1038/npp.2013.351. Epub 2014 Jan 2. PMID 24385133
- [Background] Worbe Y, Savulich G, de Wit S, Fernandez-Egea E, Robbins TW. Tryptophan Depletion Promotes Habitual over Goal-Directed Control of Appetitive Responding in Humans. Int J Neuropsychopharmacol. 2015 Feb 5;18(10):pyv013. doi: 10.1093/ijnp/pyv013. PMID 25663044
- [Background] Worbe Y, Palminteri S, Savulich G, Daw ND, Fernandez-Egea E, Robbins TW, Voon V. Valence-dependent influence of serotonin depletion on model-based choice strategy. Mol Psychiatry. 2016 May;21(5):624-9. doi: 10.1038/mp.2015.46. Epub 2015 Apr 14. PMID 25869808
- [Background] Park SB, Coull JT, McShane RH, Young AH, Sahakian BJ, Robbins TW, Cowen PJ. Tryptophan depletion in normal volunteers produces selective impairments in learning and memory. Neuropharmacology. 1994 Mar-Apr;33(3-4):575-88. doi: 10.1016/0028-3908(94)90089-2. PMID 7984295
- [Background] Sahakian BJ, Morris RG, Evenden JL, Heald A, Levy R, Philpot M, Robbins TW. A comparative study of visuospatial memory and learning in Alzheimer-type dementia and Parkinson's disease. Brain. 1988 Jun;111 ( Pt 3):695-718. doi: 10.1093/brain/111.3.695. PMID 3382917
- [Background] Bland AR, Roiser JP, Mehta MA, Schei T, Boland H, Campbell-Meiklejohn DK, Emsley RA, Munafo MR, Penton-Voak IS, Seara-Cardoso A, Viding E, Voon V, Sahakian BJ, Robbins TW, Elliott R. EMOTICOM: A Neuropsychological Test Battery to Evaluate Emotion, Motivation, Impulsivity, and Social Cognition. Front Behav Neurosci. 2016 Feb 24;10:25. doi: 10.3389/fnbeh.2016.00025. eCollection 2016. PMID 26941628
- [Derived] Armand S, Langley C, Johansen A, Ozenne B, Overgaard-Hansen O, Larsen K, Jensen PS, Knudsen GM, Sahakian BJ, Stenbaek DS, Fisher PM. Functional brain responses to emotional faces after three to five weeks of intake of escitalopram in healthy individuals: a double-blind, placebo-controlled randomised study. Sci Rep. 2024 Feb 7;14(1):3149. doi: 10.1038/s41598-024-51448-2. PMID 38326352
- [Derived] Langley C, Armand S, Luo Q, Savulich G, Segerberg T, Sondergaard A, Pedersen EB, Svart N, Overgaard-Hansen O, Johansen A, Borgsted C, Cardinal RN, Robbins TW, Stenbaek DS, Knudsen GM, Sahakian BJ. Chronic escitalopram in healthy volunteers has specific effects on reinforcement sensitivity: a double-blind, placebo-controlled semi-randomised study. Neuropsychopharmacology. 2023 Mar;48(4):664-670. doi: 10.1038/s41386-022-01523-x. Epub 2023 Jan 23. PMID 36683090